CLINICAL TRIAL: NCT05518851
Title: Treatments and Outcomes in Patients With Primary Cutaneous Lymphoma: a Nationwide Multi-center Prospective Study in China
Brief Title: TreAtments and outComes in paTients With prImary CutAneous Lymphoma
Acronym: TACTICAL
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yang WANG, Department of Dermatology and Venereology, Peking University First Hospital
Other Study IDs: PKU2022265
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Primary Cutaneous Lymphoma
Keywords: Primary Cutaneous Lymphoma; Treatment; Survival; China; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to further improve the diagnosis and treatment level of primary cutaneous lymphoma in China, the National Clinical Center for Skin and Immune Diseases established a standardized diagnosis and treatment center for primary cutaneous lymphoma to systematically and effectively understand the current treatment status of patients with primary cutaneous lymphoma, as well as the efficacy and safety of various treatment methods during practices, so as to further improve the diagnosis and treatment level of primary cutaneous lymphoma and help patients with primary cutaneous lymphoma.

DETAILED DESCRIPTION:
Primary cutaneous lymphomas (PCLs) are defined as non-Hodgkin lymphomas presenting in the skin with no evidence of extracutaneous disease at the time of diagnosis. Primary cutaneous lymphomas include a heterogeneous group of cutaneous T-cell lymphomas (CTCLs) and cutaneous B-cell lymphomas (CBCLs). The different types of PCLs have highly characteristic clinical and histologic features, often a completely different clinical behavior and prognosis, and require a different type of treatment. Various studied in terms of the treatment and outcome of patients with different types of PCLs has been conducted in recent years. While the data of Chinese patients with PCLs are limited. Considering the different proportion of PCLs and limited treatment modalities in China, a nationwide multi-center prospective study is designed to summarize the current treatment status and outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the participatin medical centers that has passed the data review of the National Clinical Center for Skin and Immune Diseases.
* Patients with a definitive pathological diagnosis of primary cutaneous lymphoma by skin biopsy.

Exclusion Criteria:

* Patients who fail to provide informed consent form.
* Patients who cannot complete the questionnaire independently or under the guidance of investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective study will span over 10 years from enrollment to follow-up data collection. Recruitment for this study will occur in the medical clinic at each participating site. Patients with primary cutaneous lymphoma will be identified at participating medical units and these patients will be invited to participate in this study. The skin biopsy will be reviewed by at least two pathologists to confirm the diagnosis. After signing the institutional review board (IRB) approved informed consent, patients will be enrolled in the study and all intend data will be collected at baseline and each scheduled follow-up time.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2032-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Type of significant therapies | At time of initiation of first significant treatment and at the each scheduled follow-up visit, through study completion, an average of 3 months
  The "significant therapies" of primary cutaneous lymphoma includes all topical and systemic therapies, radiotherapy, or phototherapy.
Duration of significant therapies | At time of initiation of first significant treatment and at the each scheduled follow-up visit, through study completion, an average of 3 months
  The "significant therapies" of primary cutaneous lymphoma includes all topical and systemic therapies, radiotherapy, or phototherapy. Recorded as "month".
Clinical response to significant therapies | At the each scheduled follow-up visit through study completion, an average of 3 months
  Clinical response are assessed by consensus response criteria in PCLs (Olsen, Elise A et al. "Primary cutaneous lymphoma: recommendations for clinical trial design and staging update from the ISCL, USCLC, and EORTC." Blood vol. 140,5 (2022): 419-437. ), recorded as "CR", "PR", "SD" or "PD".
Objective response rate(ORR) | Through study completion, an average of 1 year.
  Proportion of patients with CR and PR.
Time-to-next treatment (TTNT) | At the time of treatment change, through study completion, an average of 3 months.
  Date of initiation of primary treatment to date of new significant treatment.
Time to response (TTR) | At the time of response, through study completion, an average of 3 months.
  Date of initiation of treatment to date when criteria for response (PR or CR) first met.
Time to treatment failure (TTF) | At the time of treatment failure, through study completion, an average of 3 months.
  Date of initiation of treatment until abandonment of therapy, causes of abandonment of therapy may include inadequate response to therapy, intolerable side effects or toxicity, disease progression, and patient withdrawal for whatever reason.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline and at time of occurrence of death, through study completion, an average of 1 year.
  Date of diagnosis to death from any cause.
Progression Free Survival (PFS) | Baseline and the time of occurrence of PD or death as a result of any cause, through study completion, an average of 1 year.
  Date of diagnosis to first date meets criteria for PD or death as a result of any cause
Disease Specific Survival (DSS) | Baseline and the time of death due to disease, through study completion, an average of 1 year.
  Date of diagnosis to death as a result of disease
Disease Free Survival (DFS) | Date when criteria for CR first met and date when criteria for relapse/recurrence or or death from any cause, through study completion, an average of 1 year.
  Date when criteria for CR first met until time of relapse/recurrence (if global CR, recurrence of disease in any one category) or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yang Wang, MD, Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - SUN YAI-SEN Memorial Hospital, SUN YAI-SEN University, Guandong, Guangdong
  - Hospital for Skin Disease, Institute of Dermatology, Chinese Academy of Medical Sciences, Peking Union Medical College, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared within the participating medical units in the study, including study protocol, informed consent form, clinical study report and statistical analysis plan. Any other institutes requesting for IPD needs to be reviewed by the National Clinical Center for Skin and Immune Diseases in China.

REFERENCES:
- [Background] Olsen EA, Whittaker S, Willemze R, Pinter-Brown L, Foss F, Geskin L, Schwartz L, Horwitz S, Guitart J, Zic J, Kim YH, Wood GS, Duvic M, Ai W, Girardi M, Gru A, Guenova E, Hodak E, Hoppe R, Kempf W, Kim E, Lechowicz MJ, Ortiz-Romero P, Papadavid E, Quaglino P, Pittelkow M, Prince HM, Sanches JA, Sugaya M, Vermeer M, Zain J, Knobler R, Stadler R, Bagot M, Scarisbrick J. Primary cutaneous lymphoma: recommendations for clinical trial design and staging update from the ISCL, USCLC, and EORTC. Blood. 2022 Aug 4;140(5):419-437. doi: 10.1182/blood.2021012057. PMID 34758074
- [Background] Willemze R, Jaffe ES, Burg G, Cerroni L, Berti E, Swerdlow SH, Ralfkiaer E, Chimenti S, Diaz-Perez JL, Duncan LM, Grange F, Harris NL, Kempf W, Kerl H, Kurrer M, Knobler R, Pimpinelli N, Sander C, Santucci M, Sterry W, Vermeer MH, Wechsler J, Whittaker S, Meijer CJ. WHO-EORTC classification for cutaneous lymphomas. Blood. 2005 May 15;105(10):3768-85. doi: 10.1182/blood-2004-09-3502. Epub 2005 Feb 3. PMID 15692063
- [Background] Willemze R, Cerroni L, Kempf W, Berti E, Facchetti F, Swerdlow SH, Jaffe ES. The 2018 update of the WHO-EORTC classification for primary cutaneous lymphomas. Blood. 2019 Apr 18;133(16):1703-1714. doi: 10.1182/blood-2018-11-881268. Epub 2019 Jan 11. PMID 30635287
- [Background] Olsen E, Vonderheid E, Pimpinelli N, Willemze R, Kim Y, Knobler R, Zackheim H, Duvic M, Estrach T, Lamberg S, Wood G, Dummer R, Ranki A, Burg G, Heald P, Pittelkow M, Bernengo MG, Sterry W, Laroche L, Trautinger F, Whittaker S; ISCL/EORTC. Revisions to the staging and classification of mycosis fungoides and Sezary syndrome: a proposal of the International Society for Cutaneous Lymphomas (ISCL) and the cutaneous lymphoma task force of the European Organization of Research and Treatment of Cancer (EORTC). Blood. 2007 Sep 15;110(6):1713-22. doi: 10.1182/blood-2007-03-055749. Epub 2007 May 31. PMID 17540844
- [Background] Jawed SI, Myskowski PL, Horwitz S, Moskowitz A, Querfeld C. Primary cutaneous T-cell lymphoma (mycosis fungoides and Sezary syndrome): part II. Prognosis, management, and future directions. J Am Acad Dermatol. 2014 Feb;70(2):223.e1-17; quiz 240-2. doi: 10.1016/j.jaad.2013.08.033. PMID 24438970
- [Background] Jawed SI, Myskowski PL, Horwitz S, Moskowitz A, Querfeld C. Primary cutaneous T-cell lymphoma (mycosis fungoides and Sezary syndrome): part I. Diagnosis: clinical and histopathologic features and new molecular and biologic markers. J Am Acad Dermatol. 2014 Feb;70(2):205.e1-16; quiz 221-2. doi: 10.1016/j.jaad.2013.07.049. PMID 24438969